CLINICAL TRIAL: NCT06911099
Title: Assessment of Transcatheter Edge-to-Edge Repair in Atrial Functional Mitral Regurgitation
Brief Title: Assessment of Transcatheter Edge-to-Edge Repair in Atrial Functional Mitral Regurgitation (ATRIAL-MR)
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Philipp von Stein, MD, University Hospital of Cologne
Other Study IDs: 24-1121
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Atrial Functional Mitral Regurgitation; Mitral Insufficiency
Keywords: atrial functional mitral regurgitation; AFMR; atrial secondary mitral regurgitation; ASMR; mitral valve transcatheter edge-to-edge repair; M-TEER
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Mitral Valve Transcatheter Edge-to-Edge Repair (M-TEER): Patients who underwent mitral valve transcatheter edge-to-edge repair. All devices may be included.
- Guideline Directed Medical Therapy: Patients who underwent conservative management with guideline directed medical therapy.
- Transcatheter Mitral Valve Replacement (TMVR): Patients who underwent transcatheter mitral valve replacement. All devices may be included.

SUMMARY:
This investigator-initiated, multicenter, international, retrospective registry aims to investigate outcomes of patients with atrial functional mitral regurgitation, as treated in clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* functional mitral regurgitation
* left ventricular ejection fraction ≥50%

Exclusion Criteria:

* age under 18 years
* known regional wall movement disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study aimes to include all patients with clinically significant mitral regurgitation of the atrial functional mitral regurgitation subtype, irrespective of the subsequent therapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality and heart-failure related rehospitalitzation | 12 months

SECONDARY OUTCOMES:
Residual Mitral Regurgitation ≤1+ | 12 months
  Rate of patients achieving residual mitral regurgitation ≤1+ measured by transthoracic echocardiography. Assessment of mitral regurgitation severity according to current guidelines (ESC/EACTS and ACC/AHA) for valvular heart disease.
All-cause mortality | 12 months
Cardiovascular mortality | 12 months
Heart failure related rehospitalization | 12 months
  Incidence of new-onset or worsening signs and symptoms of heart failure that required urgent therapy and resulted in hospitalization.
Unplanned mitral valve intervention | 12 months
  Incidence of unplanned surgical or transcatheter re-intervention, heart transplantation or left ventricular assist device implantation.
New York Heart Association (NYHA) class III or IV | 12 months
  Assessment of New York Heart Association (NYHA) classification stage (in- or outpatient), with the minimum of I (no symptoms) and the maximum of IV (dyspnea at rest), with higher values indicating worse functional capacity.
6 Minute Walking Distance | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christos Iliadis, MD, Principal Investigator — Heart Center, Department III of Internal Medicine, Faculty of Medicine and University Hospital Cologne, University of Cologne, Kerpener Straße 62, 50937, Cologne, Germany
Locations (22):
- Montefiore Medical Center, The Bronx, New York, United States
- St. Michael's Hospital, Toronto, Canada
- France (2):
  - Bordeaux University Hospital, Bordeaux
  - University Hospital Center of Nantes, Nantes
- Germany (10):
  - LMU Klinikum, Munich, Bavaria
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - HDZ Bad Oeynhausen, Bad Oeynhausen
  - Heart Center Bonn, Bonn
  - University Hospital of Düsseldorf, Düsseldorf
  - University Heart and Vascular Center Hamburg, Hamburg
  - University Hospital Schleswig-Holstein, Kiel
  - Heart Center Leipzig at University of Leipzig, Leipzig
  - Heart Center of the University Medical Center Mainz, Mainz
  - University Heart Center Ulm, Ulm
- Italy (3):
  - University of Brescia, Brescia
  - San Raffaele University Hospital, Milan
  - University of Pisa, Pisa
- Spain (5):
  - Hospital Clinic of Barcelona, Barcelona
  - Reina Sofia University Hospital, Córdoba
  - University Hospital of León, León
  - Asturias Central University Hospital, Oviedo
  - University Hospital Alvaro Cunqueiro, Vigo